CLINICAL TRIAL: NCT03791502
Title: Effect of Different Volumes of Training of Pilates Exercises on Muscle Strength, Postural Balance, Flexibility, Functional Autonomy, Depressive Symptoms and Pulmonary Function on Elderly
Brief Title: Effect of Different Volumes of Training of Pilates Exercises on Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Mônica Batista Duarte Caetano, Postgraduate Student of the Post-graduation Program in Rehabilitation Sciences da University de Brasilia, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MP2018
Record Dates: First submitted 2018-11-07; First posted 2019-01-02 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Aging; Exercise Movement Techniques
Keywords: Exercise Movement Techniques; Elderly; Muscular Strength; Postural Balance; Flexibility; Pilates

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into three groups, two intervention groups and one group will be the control. The randomization process will be done by a person who does not participate in the survey, at random.org, and concealment of the allocation will occur using opaque and sealed envelopes.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates Method Exercises - lower volume (Experimental): The prescription will consist of 18 exercises, performed in a single series of seven to 10 repetitions, 60 seconds rest between exercises. Each week the exercises will be changed and the same exercise can only be repeated every three weeks. The progression will occur increasing the resistance of the springs and the level of difficulty of the exercises, but without modifying the repetitions. Training intensity will be measured using Modified Borg's Perceived Effort Scale and then kept moderate throughout the program.
  Interventions: Other: Pilates Method Exercises
- Pilates Method Exercises - higher volume (Experimental): The participants will conduct a Pilates exercise program based on the recommendations of the American College Medicine of Sports. The prescription will consist of 12 exercises, performed in three sets of seven to ten repetitions and 60s of rest between sets. Every four weeks the exercises will be changed. The progression will occur increasing the resistance of the springs and the level of difficulty of the exercises. Training intensity will be measured using Modified Borg's Perceived Effort Scale and then kept moderate throughout the program.
  Interventions: Other: Pilates Method Exercises
- Group control (No Intervention): The subjects allocated in the control group will remain with their usual activities, and after the reevaluation will be offered the intervention that presents the greater size of effect.

INTERVENTIONS:
Other: Pilates Method Exercises — Pilates Method exercises performed on the apparatus, on the ground and with accessories. They will always be performed by a physiotherapist with teaching certification in the Pilates methodology and will be supervised by two properly trained physiotherapy trainees. Participants will start the exercise program in small groups of up to 8 people, twice a week for 60 minutes, for 12 weeks, totaling 24 sessions. The first day of intervention for both groups will be devoted to explaining the six principles described by Joseph Pilates: centralization, concentration, control, precision, fluidity and breathing, and some fundamentals such as the neutral position of the spine. And in all sessions, these principles will be remembered by the physiotherapist.
  Arms: Pilates Method Exercises - higher volume; Pilates Method Exercises - lower volume

SUMMARY:
It will be an experimental study conducted with elderly of both sexes, these will be divided randomly into three groups and the intervention will happen twice a week, for 60 minutes, for 12 weeks. The aim of the study is to compare the effect of different volumes of Pilates exercise training on muscle strength, postural balance, flexibility, functional autonomy, depressive symptoms and lung function in the elderly community. The investigators believe that Pilates exercises will have beneficial effects for the elderly, but the hypothesis is that the group that performs a greater volume of Pilates exercise training will have a greater improvement in the investigated outcomes than the group with the lowest volume.

DETAILED DESCRIPTION:
Aging is an involuntary and progressive process that leads to biological, structural and functional changes such as loss of mass and muscle strength. The aging process leads to changes in the visual, vestibular, sensory and motor systems, causing slow reaction time, compromising the postural balance. Flexibility and mobility also tend to decrease with aging favoring the onset of lesions and loss of functional autonomy. The regular practice of physical exercise helps to prevent these changes related to aging. Among the various possibilities of physical exercise, the Pilates method has been well-suited for the elderly, since it incorporates the training components recommended by the American College of Sports Medicine (ACSM), is the strength, balance, and flexibility. However, researchers have questioned the lack of scientific evidence that confirms all the benefits of the method, especially in the elderly. The findings described in the literature are still controversial. A systematic review of six randomized controlled trials (RCTs) has shown limited evidence in improving strength, flexibility, and balance in both sexes.

Physical decline negatively affects the personal autonomy and quality of life of the elderly and Pilates seems to have positive effects on these aspects. Rodrigues et al. (2010) observed a significant evolution in the functional performance of healthy elderly women in rising from the seated position (11.8%) and lying position (26%) and a significant improvement in quality of life (p = 0.04) after intervention with Pilates exercises . As for depressive symptoms, Mokhtari et al. (2013) identified a significant reduction (p <0.007) in this symptomatology after Pilates practice. However, both studies reached only two points on the PEDro Scale. Recent investigations found a significant increase in maximal inspiratory pressure (MIP) of 19.5%, maximal expiratory pressure (MEP) of 8.7% and Abdominal Transversal thickness of 42.3% after the program. However, the study presented some limitations, such as the absence of a control group and the inability of the blindness of the evaluators.

It is also important to highlight the lack of reports on how the programs are carried out and when there is a description there is a heterogeneity in the prescription of the exercises. In the two reviews cited above, only two of the included studies presented the prescribed volume: ten replicates and three series of ten repetitions. Some studies have also described the volume: two sets of ten repetitions, two to four sets of 15 to 20 seconds of contraction for isometric exercises and 15 to 20 repetitions for dynamic exercises. A single series of 10 replicates with a 30-second interval between the series. It is known that the literature suggests for the muscular strength gain in the elderly a training volume of two to three sets per exercise, seven to ten repetitions per set and a moderate to high intensity and as noted most Pilates exercise programs have not followed these recommendations. The aim of the study is to compare the effect of different volumes of Pilates exercise training on muscle strength, postural balance, flexibility, functional autonomy, depressive symptoms and lung function in the elderly community.

The elderly will be invited through advertisements in social networks, local media, and posters distributed in the centers for the coexistence of the elderly, health centers and churches. Initially, each individual who agrees to participate in the study will sign the Free and Informed Consent Form. Next, the investigators will collect the data referring to the variables: cognitive aptitude, sociodemographic, clinical characterization, and anthropometric measurements. All participants will be evaluated for muscle strength, balance, flexibility, functional autonomy, depression and lung function before and after the intervention, including those who do not complete 80% of their presence during the intervention period. For the self-report questionnaires an evaluator will be trained and for the performance questionnaires/tests two evaluators will be trained and they will be blind to the intervention.

The risks of participating in the research are: the participants feel embarrassed in some interview questions, present some imbalance and risk of falls, muscle aches and increased blood pressure (BP) and heart rate (HR). However, to minimize them, the participant may refuse to answer any of the questions and interrupt the interview, as each position of the balance tests the interviewer will first demonstrate the task, then support the participants and only withdraw support after the consent of the participant, always standing next to it. The stretching will be performed in case of muscle discomfort and the monitoring of cardiorespiratory variables will be done.

How much of the benefits will participants be contributing to a greater knowledge about the effects of Pilates exercises in the elderly, the results obtained with the research will favor the formulation of adequate exercise programs and an improvement of care for the elderly, improving the quality of care, in the prevention of functional problems and falls. In addition, participants will have a thorough assessment of their overall health, well-being, and physical and functional aspects and may improve the deficiencies presented by performing Pilates exercises. Pilates will promote improved strength, muscular flexibility and well-being and provide socialization.

ELIGIBILITY:
Inclusion Criteria:

* To present cognitive aptitude according to the Mental State Mini-Exam (MMSE)
* Independent walking, without the use of auxiliary walking devices;
* Not participating in other physical intervention research;
* Not having undergone physiotherapeutic treatment and not having participated in a structured physical activity in the previous month;
* Do not present neurological diseases, history of fractures or recent surgeries and serious cardiorespiratory diseases.

Exclusion Criteria:

* Failure to attend all stages of evaluation;
* They did not complete 80% of the intervention;

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength of lower limbs | 12 weeks
  The Biofeedback System will be used for the practice of resistance exercises with elastic overload (E-lastic®). E-lastic® will measure maximal isometric voluntary contraction of the knee flexor and extensor muscles, flexors, extensors, adductors and hip abductors before and after the intervention. For the acquisition of force signals, a load cell is used to provide an electrical signal proportional to the force that deforms the equipment. The participants will perform 3 repetitions, maintaining the contraction for 5 seconds, with 60 seconds of recovery and the highest value will be recorded.
change in muscle strength and resistance of lower limbs | 12 weeks
  The 30-second chair stand test (30-s CST) will be used. It consists of getting up and sitting on a chair as many times as possible within 30 seconds. A seat with backrest and without armrest (with a seat height of 45 cm) is used. Initially, participants remain seated and are instructed to look forward after command "1, 2, 3, will" they raise with their arms crossed on their chest. The evaluator will explain and demonstrate the test and the participant will do once for familiarization. You will be given a rest of 2 minutes to start the test.
Change in palmar grip strength | 12 weeks
  Will be measured using the Saehan® hydraulic palmar gripper dynamometer, the position recommended by the American Society of Hand Therapists (ASHT) will be adopted: sitting comfortably positioned with shoulder lightly bent, elbow bent at 90 °, forearm in neutral position and, finally, the position of the handle may vary from 0 ° to 30 ° of extension. It will be used to record the maximum and average manual grip strength of three measurements and the values will be compared with the reference values.
Change in static postural balance | 12 weeks
  The static balance will be evaluated by measuring the time each participant can maintain in three progressively more difficult positions: semi-tandem, tandem and unipedal support. In all positions the individuals must be with their hands on their waist, the total time to stay in each position is 30 seconds and it will have 3 attempts in each position and the best time will be recorded. The evaluator will demonstrate the test once.
Change in dynamic postural balance (TUG) | 12 weeks
  To evaluate the dynamic balance, the Timed Up and Go Test (TUG) will be used. The TUG starts with the participant sitting in the chair, in the "go" command, he gets up from the chair, walks 3 meters at a comfortable pace, turns around, goes back to the chair and sits down. It will be demonstrated once and then it will do a repeat for familiarization.
Change in dynamic postural balance (Step) | 12 weeks
  To evaluate the dynamic balance, the Step Test will be used. The Alternative Step Test the participant is asked to make eight beats of foot, alternating between right and left, on a step in front of him with a height of 18 cm. Time will be timed and used in the analyzes. The test should be performed in 10 seconds.
Change in flexibility | 12 weeks
  To evaluate the flexibility of the hamstring muscles will be used the Sit and Go Test, using the Wells bench, participants will remain without footwear, sitting with knees extended, shoulders flexed, elbows extended and hands overlapped. Participants should perform trunk flexion at the front, perform a forced expiration, and move the seat ladder as far as possible, this procedure will be performed three times and immediately noted by the evaluator, with the best.

SECONDARY OUTCOMES:
Functional Autonomy | 12 weeks
  The functional autonomy of the upper limbs will be evaluated by the dressing test and a t-shirt. Initially the evaluator will explain the test and the volunteer will do a brief training with two replicates. The execution time is marked in seconds and the shorter the execution time, the better the result. The subject must make two attempts, where the best performance attempt will be recorded.
Depressive symptoms | 12 weeks
  The Geriatric Depression Scale will be used for the evaluation of depressive symptoms in the elderly and screening for depression among older people. Geriatric depression scale will be presented as an interview and the questions have a yes / no format to be easy to understand. The short version consists of 15 questions, one point is given for each "yes" answer and the number of points is added to provide a single score. The score ranges from 0 to 15 and a score of zero to five is considered normal, six to ten indicates mild depression and 11 to 15 suggests severe depression.
Change in respiratory muscle strength | 12 weeks
  Respiratory muscle strength will be measured by assessing maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) in cmH2O. These measures represent the strength of the inspiratory and expiratory muscles respectively. It will be using the manometer of the brand Globalmed® MVD300, calibrated, patient seated at 90º, a nasal clip and a nozzle connected to the equipment will be placed. In order to assess MIP, a maximum expiration up to the residual volume and, in the sequence, a maximum sustained forced inspiration will be required. And to assess PEmax inspiration will be required up to the total lung capacity and, subsequently, a forced maximum expiration up to the residual volume. Three reproducible measurements will be made, with variation less than 10% and the values found will be compared with those predicted.
Change in pulmonary function (FVC) | 12 weeks
  Pulmonary function will also be evaluated by spirometry. The test measures forced vital capacity (FVC) in liters (L). A One Flow® portable spirometer will be used, the individual will be seated with the head in the neutral position, inspiration will be requested up to the total lung capacity (CPT) and, thereafter, a maximum expiration, with an explosive start, to the residual volume (lasting at least 6 seconds). A maximum of eight replications will be performed until three reproducible measures (less than 10% difference), 60 seconds of interval between measurements, will be considered the best value. It is recommended to compare the values obtained with predicted equations
Change in pulmonary function (FEV1) | 12 weeks
  Pulmonary function will also be evaluated by spirometry. The test measures the forced expiratory volume in the first second (FEV1) in liters (L). A One Flow® portable spirometer will be used, the individual will be seated with the head in the neutral position, inspiration will be requested up to the total lung capacity (CPT) and, thereafter, a maximum expiration, with an explosive start, to the residual volume (lasting at least 6 seconds). A maximum of eight replications will be performed until three reproducible measures (less than 10% difference), 60 seconds of interval between measurements, will be considered the best value. It is recommended to compare the values obtained with predicted equations
Change in pulmonary function (FEV1 / FVC ratio) | 12 weeks
  Pulmonary function will also be evaluated by spirometry. The test measures the FEV1 / FVC ratio. A One Flow® portable spirometer will be used, the individual will be seated with the head in the neutral position, inspiration will be requested up to the total lung capacity (CPT) and, thereafter, a maximum expiration, with an explosive start, to the residual volume (lasting at least 6 seconds). A maximum of eight replications will be performed until three reproducible measures (less than 10% difference), 60 seconds of interval between measurements, will be considered the best value. It is recommended to compare the values obtained with predicted equations

CONTACTS AND LOCATIONS:
Overall Officials: Mônica D Caetano, Principal Investigator — University of Brasilia
Locations (1):
- Mônica Batista Duarte Caetano, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C; American College of Sports Medicine; American Heart Association. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1094-105. doi: 10.1161/CIRCULATIONAHA.107.185650. Epub 2007 Aug 1. PMID 17671236
- [Background] Delmonico MJ, Harris TB, Lee JS, Visser M, Nevitt M, Kritchevsky SB, Tylavsky FA, Newman AB; Health, Aging and Body Composition Study. Alternative definitions of sarcopenia, lower extremity performance, and functional impairment with aging in older men and women. J Am Geriatr Soc. 2007 May;55(5):769-74. doi: 10.1111/j.1532-5415.2007.01140.x. PMID 17493199
- [Background] Estrada M, Kleppinger A, Judge JO, Walsh SJ, Kuchel GA. Functional impact of relative versus absolute sarcopenia in healthy older women. J Am Geriatr Soc. 2007 Nov;55(11):1712-9. doi: 10.1111/j.1532-5415.2007.01436.x. PMID 17979895
- [Background] Sturnieks DL, St George R, Lord SR. Balance disorders in the elderly. Neurophysiol Clin. 2008 Dec;38(6):467-78. doi: 10.1016/j.neucli.2008.09.001. Epub 2008 Oct 7. PMID 19026966
- [Background] Milanovic Z, Pantelic S, Trajkovic N, Sporis G, Kostic R, James N. Age-related decrease in physical activity and functional fitness among elderly men and women. Clin Interv Aging. 2013;8:549-56. doi: 10.2147/CIA.S44112. Epub 2013 May 21. PMID 23723694
- [Background] Stathokostas L, McDonald MW, Little RM, Paterson DH. Flexibility of older adults aged 55-86 years and the influence of physical activity. J Aging Res. 2013;2013:743843. doi: 10.1155/2013/743843. Epub 2013 Jun 19. PMID 23862064
- [Background] de Oliveira Francisco C, de Almeida Fagundes A, Gorges B. Effects of Pilates method in elderly people: Systematic review of randomized controlled trials. J Bodyw Mov Ther. 2015 Jul;19(3):500-8. doi: 10.1016/j.jbmt.2015.03.003. Epub 2015 Mar 20. PMID 26118523
- [Background] Irez GB, Ozdemir RA, Evin R, Irez SG, Korkusuz F. Integrating pilates exercise into an exercise program for 65+ year-old women to reduce falls. J Sports Sci Med. 2011 Mar 1;10(1):105-11. eCollection 2011. PMID 24149302
- [Background] Bullo V, Bergamin M, Gobbo S, Sieverdes JC, Zaccaria M, Neunhaeuserer D, Ermolao A. The effects of Pilates exercise training on physical fitness and wellbeing in the elderly: A systematic review for future exercise prescription. Prev Med. 2015 Jun;75:1-11. doi: 10.1016/j.ypmed.2015.03.002. Epub 2015 Mar 12. PMID 25773473
- [Background] Siqueira Rodrigues BG, Ali Cader S, Bento Torres NV, Oliveira EM, Martin Dantas EH. Pilates method in personal autonomy, static balance and quality of life of elderly females. J Bodyw Mov Ther. 2010 Apr;14(2):195-202. doi: 10.1016/j.jbmt.2009.12.005. Epub 2010 Jan 29. PMID 20226367
- [Background] Mallery LH, MacDonald EA, Hubley-Kozey CL, Earl ME, Rockwood K, MacKnight C. The feasibility of performing resistance exercise with acutely ill hospitalized older adults. BMC Geriatr. 2003 Oct 7;3:3. doi: 10.1186/1471-2318-3-3. PMID 14531932
- [Background] Bergamin M, Gobbo S, Bullo V, Zanotto T, Vendramin B, Duregon F, Cugusi L, Camozzi V, Zaccaria M, Neunhaeuserer D, Ermolao A. Effects of a Pilates exercise program on muscle strength, postural control and body composition: results from a pilot study in a group of post-menopausal women. Age (Dordr). 2015 Dec;37(6):118. doi: 10.1007/s11357-015-9852-3. Epub 2015 Nov 15. PMID 26578458
- [Background] Markovic G, Sarabon N, Greblo Z, Krizanic V. Effects of feedback-based balance and core resistance training vs. Pilates training on balance and muscle function in older women: a randomized-controlled trial. Arch Gerontol Geriatr. 2015 Sep-Oct;61(2):117-23. doi: 10.1016/j.archger.2015.05.009. Epub 2015 May 27. PMID 26036209
- [Background] Oliveira LC, Pires-Oliveira DA, Abucarub AC, Oliveira LS, Oliveira RG. Pilates increases isokinetic muscular strength of the elbow flexor and extensor muscles of older women: A randomized controlled clinical trial. J Bodyw Mov Ther. 2017 Jan;21(1):2-10. doi: 10.1016/j.jbmt.2016.03.002. Epub 2016 Mar 10. PMID 28167180
- [Background] Borde R, Hortobagyi T, Granacher U. Dose-Response Relationships of Resistance Training in Healthy Old Adults: A Systematic Review and Meta-Analysis. Sports Med. 2015 Dec;45(12):1693-720. doi: 10.1007/s40279-015-0385-9. PMID 26420238
- [Background] Neri AL, Ongaratto LL, Yassuda MS. Mini-Mental State Examination sentence writing among community-dwelling elderly adults in Brazil: text fluency and grammar complexity. Int Psychogeriatr. 2012 Nov;24(11):1732-7. doi: 10.1017/S104161021200097X. Epub 2012 Jul 5. PMID 22874587
- [Background] Barker AL, Talevski J, Bohensky MA, Brand CA, Cameron PA, Morello RT. Feasibility of Pilates exercise to decrease falls risk: a pilot randomized controlled trial in community-dwelling older people. Clin Rehabil. 2016 Oct;30(10):984-996. doi: 10.1177/0269215515606197. Epub 2015 Sep 18. PMID 26385357
- [Background] Bird ML, Fell J. Positive long-term effects of Pilates exercise on the aged-related decline in balance and strength in older, community-dwelling men and women. J Aging Phys Act. 2014 Jul;22(3):342-7. doi: 10.1123/japa.2013-0006. Epub 2013 Aug 6. PMID 23921206
- [Background] Oliveira LC, Oliveira RG, Pires-Oliveira DA. Comparison between static stretching and the Pilates method on the flexibility of older women. J Bodyw Mov Ther. 2016 Oct;20(4):800-806. doi: 10.1016/j.jbmt.2016.01.008. Epub 2016 Feb 3. PMID 27814860
- [Background] Lord SR, Menz HB, Tiedemann A. A physiological profile approach to falls risk assessment and prevention. Phys Ther. 2003 Mar;83(3):237-52. PMID 12620088
- [Background] McCarthy EK, Horvat MA, Holtsberg PA, Wisenbaker JM. Repeated chair stands as a measure of lower limb strength in sexagenarian women. J Gerontol A Biol Sci Med Sci. 2004 Nov;59(11):1207-12. doi: 10.1093/gerona/59.11.1207. PMID 15602077
- [Background] Wells C, Kolt GS, Bialocerkowski A. Defining Pilates exercise: a systematic review. Complement Ther Med. 2012 Aug;20(4):253-62. doi: 10.1016/j.ctim.2012.02.005. Epub 2012 Mar 13. PMID 22579438

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT03791502/Prot_SAP_001.pdf